CLINICAL TRIAL: NCT05406349
Title: Neural Mechanisms of Spatial Representations Beyond the Self
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Matthias Stangl, Principal Investigator, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 7450E; R00NS126715 (NIH)
Record Dates: First submitted 2022-05-25; First posted 2022-06-06 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy Intractable
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Electrophysiological recordings in participants with intracranially implanted electrodes (Other): All participants will perform behavioral tasks that test their spatial navigation and memory performance in self-navigation and observation tasks.
  Interventions: Behavioral: Self-navigation task; Behavioral: Observation task

INTERVENTIONS:
Behavioral: Self-navigation task — Participants will perform a self-navigation task with two experimental conditions: Either they will be asked to walk towards a visible wall-mounted sign, or they will be asked to find and learn a hidden target location within the experimental room.
Behavioral: Observation task — Participants will sit on a chair in a corner of the room (RNS participants) or watch a video that was recorded from the corner of the room (EMU participants). They will be asked to keep track of another person's location who is walking around the room, and to press a button whenever the other person crosses a previously-learned target location.

SUMMARY:
Spatial navigation is a fundamental human behavior, and deficits in navigational functions are among the hallmark symptoms of severe neurological disorders such as Alzheimer's disease. Understanding how the human brain processes and encodes spatial information is thus of critical importance for the development of therapies for affected patients. Previous studies have shown that the brain forms neural representations of spatial information, via spatially-tuned activity of single neurons (e.g., place cells, grid cells, or head direction cells), and by the coordinated oscillatory activity of cell populations. The vast majority of these studies have focused on the encoding of self-related spatial information, such as one's own location, orientation, and movements. However, everyday tasks in social settings require the encoding of spatial information not only for oneself, but also for other people in the environment. At present, it is largely unknown how the human brain accomplishes this important function, and how aspects of human cognition may affect these spatial encoding mechanisms. This project therefore aims to elucidate the neural mechanisms that underlie the encoding of spatial information and awareness of others. Specifically, the proposed research plan will determine how human deep brain oscillations and single-neuron activity allow us to keep track of other individuals as they move through our environment. Next, the project will determine whether these spatial encoding mechanisms are specific to the encoding of another person, or whether they can be used more flexibly to support the encoding of moving inanimate objects and even more abstract cognitive functions such as imagined navigation. Finally, the project will determine how spatial information is encoded in more complex real-world scenarios, when multiple information sources (e.g., multiple people) are present. To address these questions, intracranial medial temporal lobe activity will be recorded from two rare participant groups: (1) Participants with permanently implanted depth electrodes for the treatment of focal epilepsy through responsive neurostimulation (RNS), who provide a unique opportunity to record deep brain oscillations during free movement and naturalistic behavior; and (2) hospitalized epilepsy patients with temporarily implanted intracranial electrodes in the epilepsy monitoring unit (EMU), from whom joint oscillatory and single-neuron activity can be recorded.

DETAILED DESCRIPTION:
This research study is based upon a unique opportunity to work with neurosurgical patients, who already have electrodes implanted in deep brain structures for clinical reasons (i.e., for the monitoring and treatment of pharmaco-resistant epilepsy). Research procedures will only be performed with patients who already have such electrodes implanted for clinical reasons; no electrodes will be implanted for research purposes, and the researchers will not have any influence on the implantation procedures of these electrodes. Two groups of participants will be asked to participate in the research study: 1. Hospitalized patients who have electrodes implanted temporarily (typically for up to two weeks) for epilepsy monitoring in the epilepsy monitoring unit (EMU participants). 2. Patients who have chronically/permanently implanted electrodes as part of the NeuroPace RNS System for the treatment of epilepsy (RNS participants). Independent from and prior to the research study, the patient's clinical care team (neurologists, neurosurgeons, etc.) decide whether electrodes or the RNS System will be implanted based solely on clinical criteria. If electrodes or the RNS System are implanted, patients will then be offered to participate in the research study; however, the decision whether or not to participate in the research study will not have any effect on the patient's treatment or clinical care.

Screening, recruitment, and consent procedures for EMU participants:

If the clinical care team decides - independent from the research study - that a patient's clinical condition merits implantation of temporary electrodes and hospitalization in the epilepsy monitoring unit (EMU), the patient's neurologists or neurosurgeons will invite the patient to participate in the research study. The neurosurgeons and neurologists make it clear to the patient that the decision to participate in the research is entirely voluntary and that the patient's medical needs will not be affected in any way by this decision. For patients who are interested in participating in the research study, the principal investigators meet with the patient to discuss the consent form. Subsequently the principal investigator also ensures that the patient fully understands the consent form and emphasizes again to the patient that participation is entirely voluntary and that the patient's decision whether to participate or not will have no effect on their medical care. If the patients are local, the research team meets with the patient at UCLA before or after pre-surgical tests. This is commonly done a 1-3 weeks before the surgery. For patients traveling long distance, the discussion may take place the day before the surgery. After discussion the patient signs the consent form to participate in the research study and it is countersigned by the principal investigator.

Screening, recruitment, and consent procedures for RNS participants:

For the proposed study, the investigators have already identified a number of patients for other ongoing studies that received NeuroPace RNS System at the UCLA medical center with RNS devices implanted in medial temporal lobe regions. These patients have been identified through their neurosurgeon or neurologist, who are part of the study team. These neurosurgeons and neurologists will inform their patients about the opportunity to participate in this research study. The neurosurgeons and neurologists make it clear to the patient that the decision to participate in the research is entirely voluntary and that the patient's medical needs will not be affected in any way by this decision. Potential subjects external to the UCLA medical center may have preliminary contact from their treating physician from a referring institution. If patients indicate interest in the study, the principal investigator, faculty sponsor, or the study coordinator will make initial direct contact via phone in a private secure location to introduce and describe the study after which further information and copy of consent form can be sent for review via secure encrypted e-mail and/or mail, if necessary. The principal investigators also ensure that the patient fully understands the consent form and emphasize again that participation is entirely voluntary and that the patient's decision whether to participate will have no effect on their medical care. Potential participants will be approached no earlier than 3 months after their RNS system placement to see if the patient would be interested in volunteering for the study. Consent may be obtained over the phone or internet for participants necessitating extended travel arrangements and accommodations. Participants, particularly those consented over the phone or via the internet, will be provided with a physical copy of the consent form and asked to sign it before performing any research procedures.

Behavioral tasks:

RNS participants will complete both freely moving and stationary view-based spatial navigation and observation tasks whereas EMU participants will complete only stationary view-based spatial navigation and observation tasks. Intracranial electroencephalographic (iEEG) activity in RNS participants, and joint single-neuron activity and local field potentials (LFP) in EMU participants will be recorded while participants complete variants of self-navigation and observation tasks, similar to our previous work. All spatial navigation and observation tasks will have the basic structure as follows:

* Self-navigation task: RNS participants will navigate an experimental room (size about 19.4 × 17.1 feet) in which 20 unique signs (combinations of a single color per wall with numbers 1 to 5) are mounted along the 4 room walls. In addition, several predefined target locations (each named with a letter) will be randomly distributed throughout the room, but not visible to participants. Participants will be repeatedly asked to navigate to one of the visible signs (e.g., "Go to sign yellow-4") or to find and learn one of the invisible target locations (e.g., "Find target location T"). EMU participants will be asked to perform the self-navigation tasks in a virtual environment, which is an exact virtual replica of the real experimental room. To ensure a maximally immersive experience, the participant will see this room from first-person perspective via a head-mounted display, and the participant will be able to virtually walk around in this room using wireless controllers. In the case of any discomfort, tasks can also be performed on a desktop computer screen.
* Observation task: RNS participants will sit in the corner of the experimental room and observe another person (i.e., an experimenter) that walks around within the room in a seemingly random trajectory (in fact, the trajectory will be pre-defined and controlled, but unknown to participants). Participants will be asked to press a button whenever the experimenter hits one of the previously-learned invisible target locations. EMU participants will also perform this task; however, EMU participants will watch the room and the other person in a video that was recorded from a corner of the room. This video will be shown in the head-mounted display, in order to mimic the experience from an observer's first-person perspective (as if the participant would actually sit in the real room corner). In the case of any discomfort, tasks can also be performed on a desktop computer screen. For different study aims, participants will be asked to perform slightly modified versions of the observation task: Instead of another person, participants will be asked to observe the movements of an inanimate object (an electric remote-controlled platform, similar to a remote-controlled toy car), or to observe not one but multiple other people that move through the experimental room. And participants will be asked to just imagine movements of other individuals and objects throughout the room, while no other individuals/objects are physically present.

Electrophysiological recordings in EMU participants during task performance:

For participants with temporarily implanted electrodes in the epilepsy monitoring unit (EMU) at UCLA, the Neuroport System (Blackrock Microsystems, Salt Lake City, UT) will be used for data acquisition, which records single-unit and LFP neuronal activity alongside the simultaneously recording clinical systems for epilepsy monitoring.

Electrophysiological recordings in RNS participants during task performance:

Participants have the chronically/permanently implanted FDA-approved RNS System for clinical reasons (i.e., treatment of epilepsy), which is designed to treat epileptic seizures by continuously recording electrophysiological activity from the patient's brain during everyday life activities, and delivering electrical stimulation when abnormal activity patterns (e.g., epileptic seizure-like activity) are detected. For the research study, the study team will use the regular recording capabilities of the RNS System, while participants perform the described navigation and memory tasks.

Motion tracking during behavioral tasks:

For RNS participants, the location of participants within the experimental room will be continuously tracked with sub-millimeter resolution using the OptiTrack motion tracking system (Natural Point Inc.). Motion tracking will not be performed for EMU participants, as these participants perform only stationary view-based tasks.

Eye tracking during behavioral tasks:

RNS participants' eye movements will be recorded using a mobile eye tracking headset, which also allows mapping of the participant's gaze (i.e., their visual focus) onto the video of an integrated 'world camera' that captures the environment from the participant's point of view. EMU participants' eye movements will be recorded with a built-in eye tracker within the head-mounted display, providing eye movement as well as gaze position data.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years of age
* Adequate visual and auditory acuity to allow neuropsychological testing
* Have undergone depth electrode placement for the purpose of epilepsy evaluation/treatment OR have NeuroPace RNS System implanted for epilepsy treatment

Exclusion Criteria:

* All DSM-V Axis I and II disorders other than nicotine-dependence
* History of brain damage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-06 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Oscillatory power | Continuous measurement during task performance on day 1 and all subsequent measurement days (up to 14 days per participant)
  It will be measured how the oscillatory power (measurement unit: microvolts-squared) of electrophysiological brain activity, as measured via intracranially implanted electrodes and an electroencephalography recording system, is modulated by task-related behavioral variables (such as the individual's spatial location, head direction, movement speed, or their distance/direction to environmental boundaries).
Oscillatory amplitude | Continuous measurement during task performance on day 1 and all subsequent measurement days (up to 14 days per participant)
  It will be measured how the oscillatory amplitude (measurement unit: microvolts) of electrophysiological brain activity, as measured via intracranially implanted electrodes and an electroencephalography recording system, is modulated by task-related behavioral variables (such as the individual's spatial location, head direction, movement speed, or their distance/direction to environmental boundaries).
Oscillatory frequency | Continuous measurement during task performance on day 1 and all subsequent measurement days (up to 14 days per participant)
  It will be measured how the frequency of an oscillation (measurement unit: Hertz), as measured via intracranially implanted electrodes and an electroencephalography recording system, is modulated by task-related behavioral variables (such as the individual's spatial location, head direction, movement speed, or their distance/direction to environmental boundaries).
Firing rate of single neurons | Continuous measurement during task performance on day 1 and all subsequent measurement days (up to 14 days per participant)
  It will be measured how the firing rate of single neurons (measurement unit: Hertz), as measured via intracranially implanted micro-electrodes and an electrophysiology recording system, is modulated by task-related behavioral variables (such as the individual's spatial location, head direction, movement speed, or their distance/direction to environmental boundaries).

OTHER OUTCOMES:
Eye movement speed | Continuous measurement during task performance on day 1 and all subsequent measurement days (up to 14 days per participant)
  It will be measured how eye movements (specifically, the speed of eye movements, quantified as changes in pupil position; measurement unit: degrees per second), as measured with a mobile eye tracking system, are modulated by task-related behavioral variables (such as the individual's spatial location, head direction, movement speed, or their distance/direction to environmental boundaries). These eye tracking data will also be used for control analyses, to test whether the primary outcome measures (electrophysiological activity change) are influenced by eye movements.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Stangl, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No